CLINICAL TRIAL: NCT03880097
Title: Enabling the Study of Metabolism in Breast Cancer Through Collection of Fresh-tissue Biopsies
Acronym: ENSEMBLE
Status: Not yet recruiting | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 17/0765
Record Dates: First submitted 2018-10-09; First posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Research Biopsy: The research biopsy is the same procedure as a standard of care percutaneous biopsy. A "core" (hollow) needle is inserted into the tumour tissue in order to collect tissue samples. The procedure is called a research biopsy as it is an additional procedure to the standard of care, used purely to collect tissue samples for research purposes.
  Interventions: Procedure: Research Biopsy

INTERVENTIONS:
Procedure: Research Biopsy — The "Research Biopsy" is a biopsy in addition to the standard of care biopsies that the patient will have to inform their diagnosis. The actual procedure is not any different to the standard per-cutaneous biopsy, this is just an additional procedure, solely for research purposes.

SUMMARY:
This study aims to evaluate how breast cancer cells metabolise nutrients in order to grow. Patients enrolled into this study will undergo a research biopsy that will aim to collect up to 4 cores of tumour tissue. These tissues will then be used in translational research to analyse how specific pro-tumorigenic events change breast cancer cell metabolism (compared to healthy cell metabolism).

DETAILED DESCRIPTION:
Comprehensive analysis linking breast tumour subtypes and their genetic profile with tumour metabolism are required. Traditional model systems are inadequate for this purpose.

1. In vitro models do not represent a true tumour environment and are a subject of prolonged adaptation to artificial cell culture conditions.
2. There is a need for in vivo and ex vivo models representing breast cancer diversity and tumour environment that can be used for predicting and testing the personalised therapies.

Metabolic analysis of fresh tissues (by metabolomics and Mass Spectrometry Imaging (MSI)) and tissues grown as patient derived xenograft models in vivo should reveal the unperturbed relationships between genetic profiles of tumour cells, tumour microenvironment and metabolic profiles of tumours. These relationships should provide new targets for metabolism-based therapies. The experimental systems required to perform this research require fresh breast cancer biopsies.

ENSEMBLE is a prospective multi-centre cohort study that aims to address these issues. Fresh breast tumour tissue will be collected from consented female participants diagnosed with invasive breast cancer, for translational research. Up to 240 participants will be enrolled over a 36-month period and clinical follow-up data will be collected for up to 5 years. Study participants will undergo a "research biopsy" (core biopsy) for translational research that aims to collect up to four cores. The procedure is the same as the standard of care percutaneous core needle biopsy that the patient will have to inform their diagnosis, however, as it is an additional procedure, it is called a "research biopsy". Wherever possible biopsy samples will be taken from the operative specimen at the time of primary surgery however, where neo-adjuvant therapy is planned in a patient's care plan, these patients will undergo a research percutaneous biopsy prior to their surgery, performed either using image-guidance or as a clinical biopsy.

Collected tumour material will be divided: a portion will immediately be frozen in liquid nitrogen, and a portion will be kept fresh. The material will be transported to the primary receiving laboratory at the Francis Crick Institute where part of the sample will be immediately engrafted into immune-deficient mice to create a patient-derived xenograft (PDX) model. The remaining primary samples and samples from PDXs will be used for genomic, metabolomic and other biochemical analyses.

Information about participant demographics, medical history and tumour characteristics will be collected at registration. Participants may be followed up for up to 5 years for clinical outcome data and to clarify information about medical history

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of newly diagnosed breast cancer
* Known ER and HER2 receptor status
* Tumour diameter ≥1cm on imaging
* Female
* Age 18 or above
* Written informed consent

Exclusion Criteria:

* Previously treated invasive breast cancer
* Primary systemic therapy for breast cancer prior to biopsy
* Oestrogen replacement therapy (HRT) within 14 days of biopsy in ER-positive tumours
* Pregnancy or breastfeeding
* Not considered suitable by clinical team

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women over the age of 18 with a new diagnosis of breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of biopsies collected | 3 years
  The primary outcome is the number of biopsies successfully collected from the 240 women approached.

SECONDARY OUTCOMES:
Breast cancer cell biology | 5 years
  Understanding how specific, pro-tumorigenic events change breast cancer cell metabolism.
Identifying vulnerabilities in breast cancer cell metabolism | 5 years
  Identifying vulnerabilities in cancer cell metabolism with a view to identification of novel therapeutic targets.

CONTACTS AND LOCATIONS:
Overall Officials: Neill Patani, MD, Principal Investigator — University College London Hospitals; Jayant Vaidya, MD, Principal Investigator — The Whittington Hospital; Michael Douek, MD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust; Amna Sherri, MD, Principal Investigator — Royal Free London NHS Foundation Trust; Laura Johnson, MD, Principal Investigator — Barts & The London NHS Trust; Robert Price, MD, Principal Investigator — King's College Hospital NHS Trust

IPD SHARING:
Plan to Share IPD: Undecided
To follow.